CLINICAL TRIAL: NCT05160285
Title: The NEVOLUTION Study: An Open Label, Single-arm, Phase II Study of Neoadjuvant Nivolumab in Locally Advanced Upper Tract Urothelial Carcinoma
Brief Title: Neoadjuvant Nivolumab for Upper Tract Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: YULISU (Other)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor-Investigator, YULISU, Assistant Professor-level Attending Physician, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCGMHCTC-2019005; CPRPG8J0011 (Other Grant/Funding Number: Chang Gung Memorial Hospital)
Record Dates: First submitted 2020-12-24; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Upper Urinary Tract Urothelial Carcinoma
Keywords: upper tract urothelial carcinoma; immune checkpoint inhibitor; neoadjuvant treatment; pathological complete response; whole exome sequencing; biomarker; RNA sequencing; ctDNA
MeSH Terms: interventions — Nivolumab; Injections

STUDY DESIGN:
Intervention Model Description: Open Label, Single-arm, Phase II Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant nivolumab treatment arm (Experimental): Nivolumab 360mg intravenous adminstration every 3 weeks
  Interventions: Drug: Nivolumab 100 MG in 10 ML Injection

INTERVENTIONS:
Drug: Nivolumab 100 MG in 10 ML Injection — If you meet all the conditions to participate in the trial, you will receive the following treatments: Your physician will give you 360 mg of Nivolumab as an intravenous infusion every 3 weeks for about 30 minutes. For safety reasons, we recommend that you stay in the hospital for 60 minutes after the initial infusion of nivolumab. There will be a total of 3 cycles of Nivolumab treatments during the study period. You will need to return every 3 weeks. Each return will collect about 50 ml (10 tsp) of blood samples, depending on local standards.

SUMMARY:
The aim of this study is to explore efficacy and safety of neoadjuvant nivolumab for non-metastatic upper tract urothelial carcinoma (UTUC), and explore the potential predictive biomarkers of immunotherapy.

DETAILED DESCRIPTION:
Upper urinary tract urothelial carcinoma (UTUC) is a malignant tumor originated from the epithelium of upper urinary tract (renal pelvis and ureter). The standard treatment of UTUC is radical nephroureterectomy with ipsilateral bladder cuff excision. For locally advanced disease, neoadjuvant chemotherapy or adjuvant chemotherapy with radiotherapy is also a considerable treatment. In general, patients with UTUC are often diagnosed in a late stage with a poor survival.

Nowadays, immune checkpoint inhibitor (ICI) emerged huge success in treatment of various type of cancers, including metastatic urothelial carcinoma. Several anti-PD1 or PD-L1 agents demonstrated an exciting response for metastatic urothelial carcinoma. The encouraging success makes clinical trials moving forward to neoadjuvant setting. In the PURE-01 study, patients with muscle-invasive bladder cancer received 3 cycles of neoadjuvant pembrolizumab achieving 39.5% pathological complete response (pCR). It brought a brand-new hope for organ-preservation treatment strategy. So far, neoadjuvant ICI has not been tested in patients with UTUC, irrespective for treatment efficacy or safety analysis. More importantly, there is still lack of reliable biomarkers to predict treatment response of ICI, which definitely an unmet medical need in clinical practice.

Therefore, the investigators proposed a phase II, open-label study of neoadjuvant nivolumab in locally advanced UTUC. Investigators believe that neoadjuvant nivolumab will achieve at least similar pCR rate compared with neoadjuvant pembrolizumab in UCB patients. Furthermore, investigators will conduct a comprehensive exploratory genomic analysis to identify the potential candidate biomarkers to predict the response of nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or clinically confirmed diagnosis of locally advanced (cT2-T4 and N0M0) urothelial carcinoma of the renal pelvis and/or ureter (UTUC). Pure urothelial carcinoma or urothelial carcinoma mixed with other histological variant are allowed, but urothelial carcinoma must be the predominant histology.
2. Have at least a measurable lesion based on RECIST 1.1 as determined by the local site investigator/radiology assessment.
3. Voluntarily agree to participate by providing written informed consent/assent for the trial.
4. Age (at the time of informed consent): 20 years and older
5. Have received no prior systemic chemotherapy for advanced urothelial carcinoma, with the following exceptions:

   1. Platinum-based chemotherapy for previous a history of ipsilateral UTUC or bladder cancer in purpose of neoadjuvant or adjuvant treatment with recurrence > 6 months from completion of therapy is permitted.
   2. Low-dose chemotherapy (e.g., low-dose cisplatin, cisplatin plus 5-FU, mitomycin plus 5-FU, or cisplatin plus paclitaxel) given concurrently with radiation to urothelial carcinoma of bladder is not considered systemic therapy.
6. Have willing to provide tissue for exploratory biomarker analysis from a newly obtained core or excisional biopsy of a tumor lesion from the renal pelvis or ureter tumor.
7. Have an ECOG PS of 0, 1, or 2.
8. Have adequate organ function as defined in Table 6. (All screening labs should be performed within 3 weeks prior to treatment initiation.)
9. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 7.5.2 - Contraception, for the course of the trial through 5 months or more after the last dose of nivolumab

Exclusion Criteria:

* 1. Is currently participating and receiving study therapy or investigational agents. Patients who withdraw of previous clinical trials should have a 4-weeks washout period of investigational drug before participating this study.

  2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to randomization.

  3. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  1. Short-term (<7 days) use of systemic corticosteroids is allowed when use is considered SOC.
  2. Subjects with vitiligo, type I diabetes mellitus, hypothyroidism, or resolved childhood asthma/atopy would be an exception to this rule.
  3. Subjects who require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the trial.

     4. Has a known additional malignancy that is progressing or requires active treatment within the past 5 years.

  <!-- -->

  1. Exceptions include basal cell carcinoma of the skin; squamous cell carcinoma of the skin that has undergone potentially curative surgery; in situ cervical cancer; early stage of prostate cancer (stage 1) with low Gleason score ≤6; and prostate-specific antigen (PSA) undetectable.
  2. A history of urothelial carcinoma, including upper tract urothelial carcinoma or bladder cancer who received curative-intent surgery (nephroureterectomy, segmentectomy, TURBT, partial cystectomy, radical cystoprostectomy) > 12 months before first-dose trial treatment will be the exception.

     5. Has a history of (non-infectious) pneumonitis or interstitial lung disease or pulmonary fibrosis diagnosed based on imaging (CT of chest preferably).

     6. Has active tuberculosis (TB) (Bacillus tuberculosis). 7. Has an active infection requiring systemic therapy within 7 days prior to the first dose of trial treatment.

     8. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 5 months or more after the last dose of nivolumab.

     9. Has a history of uncontrolled or significant cardiovascular disease meeting any of the following:

  <!-- -->

  1. Myocardial infarction within 180 days before first-dose of trial treatment
  2. New York Heart Association (NYHA) class III or IV congestive heart failure
  3. Myocarditis, no matter what etiology should be excluded
  4. Arrhythmia requiring treatment (e.g. atrial fibrillation/flutter, ventricular tachycardia or fibrillation, paroxysmal supraventricular tachycardia, symptomatic bradycardia, sick sinus syndrome or high-grade atrioventricular block).
  5. Has permanent pacemaker implantation or implantable cardioverter defibrillator (ICD).

     10. Has received prior therapy with an anti-PD-1, or anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).

     11. Has undergone major surgery (any surgery involving general anesthesia) within 28 days before first-dose of study therapy.

     12. Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).

     13. Has known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected). Controlled (treated) hepatitis B subject will be allowed if they meet the following criteria:

  <!-- -->

  1. Antiviral therapy for HBV must be given for at least 8 weeks and HBV viral load must be less than 100 IU/mL prior to first dose of study drug.
  2. Subject who are anti-HBc (+), negative for HBsAg, negative for anti-HBs and have an HBV viral load under 100 IU/mL don't need HBV anti-viral prophylaxis.

     14. Has received a live virus vaccine within 30 days of planned start of trial therapy.

     15. Has known CNS metastases and/or leptomeningeal carcinomatosis. 16. Has symptomatic ascites or pleural effusion. 17. Has had a prior allogeneic stem cell or bone marrow transplant. 18. Has received any unapproved or unlicensed drug (e.g. marketed drugs unapproved for urothelial carcinoma, investigational use of drugs, herb combination) within 28 days before first-dose of study drug.

     19. Are otherwise unfit for the study in the investigator's or sub-investigator's opinion.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-12-25 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate (pCR) | 1 month post neoadjuvant nivolumab and surgery
  determined by genitourologic pathologist

SECONDARY OUTCOMES:
Treatment related adverse effect | 3 months during nivolumab treatment
  determined by CTCAE
Surgical complication | 1 month within surgery
  determined by Clavien-Dindo classification
Objective response rate | 3 months
  determined by RECIST 1.1 criteria
Disease free survival | 6 months
  Milestone time points analysis of DFS6, DFS12, DFS 18 and median PFS by investigator assessment per RECIST 1.1
Overall survival | 6 months
  Milestone time points analysis of OS6, OS12, OS18 and median OS by investigator assessment per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Li Su, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No